CLINICAL TRIAL: NCT04272086
Title: Effect of Transversus Abdominal Plane Block Using Liposomal Bupivacaine Versus Standard Bupivacaine for Open Myomectomy: A Prospective Randomized Control Trial
Brief Title: Utility of Liposomal Bupivacaine Transversus Abdominal Plane Block for Open Myomectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Daniel Katz, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GCO 19-1807
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Fibroid Uterus
Keywords: Fibroid uterus; Myomectomy; Abdominal myomectomy
MeSH Terms: conditions — Leiomyoma | interventions — Bupivacaine; Saline Solution

STUDY DESIGN:
Intervention Model Description: Double blind randomized control trial with intervention arm as liposomal bupivacaine tap and intervention as standard bupivacaine tap
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The only people who will be unblinded are the members of the block team, who are not members of the care team nor the study team. They will open the envelopes, draw up the medications and cover the syringes with opaque paper such that no one can tell the contents.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bupivacaine TAP (Placebo Comparator): TAP block with 30 mL 0.25% bupivacaine mixed with 10 mL normal saline for a total of 40 mL per side
  Interventions: Drug: Bupivacaine; Drug: normal saline
- Liposomal bupivacaine TAP (Experimental): TAP block with 10mL liposomal bupivacaine, 20mL 0.25% bupivacaine, and 10mL normal saline for a total of 40 mL per side
  Interventions: Drug: Bupivacaine; Drug: Bupivacaine liposome; Drug: normal saline

INTERVENTIONS:
Drug: Bupivacaine — 0.25%
Drug: Bupivacaine liposome — 10mL
  Arms: Liposomal bupivacaine TAP
Drug: normal saline — 10ml

SUMMARY:
The study team will be randomizing patients presenting for open myomectomy to either received transversus abdominal plane blocks with either liposomal bupivacaine or standard bupivacaine. The study team will be analyzing the impact of local anesthetic on opiate consumption as the investigator's primary endpoint with other secondary endpoints.

DETAILED DESCRIPTION:
After consent, patients will be randomized to either liposomal bupivacaine Transversus Abdominal Plane (TAP) vs standard bupivacaine TAP. Blocks will occur post induction and pre incision. Only the block team (not the anesthesia team nor the care team) will be unblinded and they will not have any impact on the data collection. The entire care team and the patient will be blinded. A standardized anesthetic regimen will be employed followed by a prescriptive post-operative pain management plan aimed at enhanced recovery. Patients will be followed for up to 96 hours and asked about their opiate consumption, pain scores, side effects, and recovery.

ELIGIBILITY:
Inclusion Criteria:

* Not pregnant
* Weight over 50kg presenting for open myomectomy
* No history of allergy to any study medication
* No history of malignant ventricular dysrhythmia, epilepsy, seizure disorder, or chronic pain syndrome other than pain from myomas
* No history of drug or alcohol use or abuse disorder or pre-existing liver disease.

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only women have uterine fibroids
Enrollment: 140 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2025-10-28 (Actual); Study Completion 2025-10-28 (Actual)

PRIMARY OUTCOMES:
Morphine Equivalents at 72 Hours | 72 hours
  Total cumulative opiates consumed converted to morphine equivalents

SECONDARY OUTCOMES:
Morphine Equivalents at 96 Hours | 96 hours
  Total cumulative opiates consumed converted to morphine equivalents
Morphine Equivalents at 48 Hours | 48 hours
  Total cumulative opiates consumed converted to morphine equivalents
Opiate Sparing Criteria at 72 hours | 72 hours
  Composite score of minimal opiate dose and additionally scores of 0 on questions 2,3,4,5,6 on OBAS scoring scale.
  Overall Benefit of Analgesic Score (OBAS) scoring scale -total scale from 0-20, low score indicates high benefit.
Quality of Recovery at 48 hours | 48 hours
  15 question quality of recovery scale, full scale from 0-150, with lower score indicating better recovery.
Quality of Recovery at 72 hours | 72 hours
  15 question quality of recovery scale, full scale from 0-150, with lower score indicating better recovery.
Area under the curve pain scale at 96 hours | 96 hours
  Sum of pain scores at 24, 48, 72, and 96 hours. Pain scale from 0-10, with higher score indicating worst pain.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Katz, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-08-05): https://cdn.clinicaltrials.gov/large-docs/86/NCT04272086/ICF_000.pdf